CLINICAL TRIAL: NCT00575913
Title: ALEX-XL: Alfuzosin XL-Lower Urinary Tract Symptoms Efficacy and Sexuality Study
Brief Title: Alfuzosin XL Lower Urinary Tract Symptoms Efficacy and Sexuality Study
Acronym: ALEX-XL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_8935
Record Dates: First submitted 2007-12-17; First posted 2007-12-18 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-04

CONDITIONS: Prostatic Diseases
MeSH Terms: conditions — Prostatic Diseases | interventions — alfuzosin

INTERVENTIONS:
Drug: Alfuzosin — Alfuzosin 10 mg One tablet per day after evening meal
  Other Names: (Xatral XL)

SUMMARY:
To assess, under daily practice conditions, the safety profile and the efficacy of a new formulation of alfuzosin administered once daily (Xatral XL) in patients with lower urinary tract symptoms (LUTS) suggestive of benign prostatic hyperplasia (BPH).

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients suffering from lower urinary tract symptoms suggestive of BPH.

Exclusion Criteria:

* Patients requiring BPH surgery immediately or within the 12 following months:

  * Acute renal obstruction
  * Chronic renal obstruction
  * Chronic renal failure from BPH
  * Bladder stone
  * Recurrent urinary tract infection
  * Other bladder pathology such as cancer of the bladder, bladder bidiverticulum (big size)
  * Hematuria from BPH
* Patients whose urinary symptoms are satisfactorily controlled on other BPH medication ( alpha-blockers or 5 alpha-reductase)
* Patients previously not improved by an alpha1-blocker treatment
* Known hypersensitivity to alfuzosin
* History of postural hypotension or syncope
* Combination with other alpha1-blockers
* Hepatic enzyme (SGOT or/and SGPT ) > 1.5 Upper Normal Limit
* Unstable angina pectoris
* Severe concomitant condition threatening life.
* Patients who had failed treatment with finasteride (Proscar)
* Patients with neuropathic bladder.
* Patients with history of previous surgery for BPH
* Patients with high risk for prostate cancer based on the clinical judgement of the investigator

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2003-09; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
improvements in urinary symptoms and quality of life index | During all the study conduct

SECONDARY OUTCOMES:
Improvement in sexual function | During all the study conduct
Improvement in maximum flow rate (determined by uroflowmetry) | During all the study conduct
Collection of spontaneously reported adverse events | At each visit

CONTACTS AND LOCATIONS:
Overall Officials: Paibulsirijit Sompob, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bangkok, Thailand